CLINICAL TRIAL: NCT02612025
Title: Effects of Combined Resistance and Endurance Training in Pediatric Cancer Patients During Intensive Treatment Phase
Brief Title: Effects of Resistance and Endurance Training in Pediatric Cancer Patients During Intensive Treatment Phase
Acronym: MUCKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Univ.Prof.Dr.med. Joerg Faber, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mucki01
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Pediatric Oncology
MeSH Terms: interventions — Exercise

ARMS (2):
- Exercise group (Experimental): Exercise training during intensive medical treatment
  Interventions: Behavioral: Exercise Training
- Control group (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Exercise Training — Exercise training during intensive medical treatment. Training mainly composed of endurance and resistance exercises. 3 to 5 times per week for six weeks.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to determine whether combined endurance and resistance training can improve muscle strength in children and adolescents with cancer during the intensive treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Malignant Tumor
* Medical Treatment in the Center for Pediatrics, Hematology, Oncology and Hemostaseology Mainz (Germany)
* > 3 years
* Signed Informed Consent

Exclusion Criteria:

* Functional and/or cognitive limitations which limit performance during training
* Orthopedic condition which hinders to adequately participate in exercise training
* Heart failure (NYHA III-IV)
* Partial or global respiratory failure
* Symptomatic coronary disease
* Serious therapy-refractory hypertonia
* Sustainable thrombocytopenia <10.000/µl, f. ex. therapy-refractory autoimmune thrombocytopenia
* Hereditary or acquired thrombocytopenia or coagulation disturbance
* Uncontrolled cerebral spasm
* CNS metastases
* Medical or psychological condition which does in the doctors opinion not allow participation in sport activity

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Muscle strength: lower limb | Six weeks (pre-post intervention)
  Lower limb muscle strength measured by the load (kg) sustained in one repetition maximum test

SECONDARY OUTCOMES:
Muscle strength: upper limb | Six weeks (pre-post intervention)
  Upper limb muscle strength measured by the load (kg) sustained in one repetition maximum test
Biomarker in Blood | At the beginning of the intervention and three and six weeks after the beginning. Comparing the two time points inbetween study groups
  Immune status and metabolic status
Body composition | Six weeks (pre-post intervention)
  Bioelectrical Impedance Analysis
Six-minute-walk performance | Six weeks (pre-post intervention)
Fatigue | six weeks (pre-post intervention)
  Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale
Quality of Life | Six weeks (pre-post intervention)
  KINDL: health related quality of life questionnaire
Cardiorespiratory performance | Six weeks (pre-post intervention)
  Ergospirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes-Gutenberg-University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Winker M, Stossel S, Neu MA, Lehmann N, El Malki K, Paret C, Joisten N, Bloch W, Zimmer P, Faber J. Exercise reduces systemic immune inflammation index (SII) in childhood cancer patients. Support Care Cancer. 2022 Apr;30(4):2905-2908. doi: 10.1007/s00520-021-06719-3. Epub 2021 Dec 3. PMID 34860287
- [Derived] Stossel S, Neu MA, Wingerter A, Bloch W, Zimmer P, Paret C, Malki KE, Baumann FT, Russo A, Henninger N, Lehmann N, Otto H, Faber J. Benefits of Exercise Training for Children and Adolescents Undergoing Cancer Treatment: Results From the Randomized Controlled MUCKI Trial. Front Pediatr. 2020 Jun 5;8:243. doi: 10.3389/fped.2020.00243. eCollection 2020. PMID 32582585